CLINICAL TRIAL: NCT06626048
Title: Optimizing an Integrated Mind and Body Treatment for Insomnia: The SLEEPS Study
Acronym: SLEEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-41821 A; R34AT012767-01 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Insomnia Disorder
Keywords: Passive Body Heating; Cognitive Behavioral Therapy for Insomnia; CBT-I; Mood Disorders; Insomnia Disorder; Digital Intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (CBT-I) and Passive Body Heating (PBH) (Experimental): Participants will receive both digital Cognitive Behavioral Therapy for Insomnia (CBT-I) and Passive Body Heating (PBH) using a sauna blanket.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Device: Passive Body Heating (PBH)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Digital cognitive behavioral therapy for insomnia (CBT-I) is a behavioral (psychotherapeutic) intervention for insomnia disorder. Participants will complete digital CBT-I online using the Sleep Healthy Using the Internet (SHUTi) program.
Device: Passive Body Heating (PBH) — Passive body heating (PBH) is a body-based treatment that participants will complete using a sauna blanket, which is similar in form factor to an adult-sized sleeping bag (head is not within the heated area). Participants will complete at least three 15-minute PBH sessions per week. Participants will complete PBH sessions in the sauna blanket placed on the floor or on a couch (i.e., not in their bed) at a setting of Level 6, 1-2 hours before bed.

SUMMARY:
This single-arm feasibility trial will provide digital cognitive behavioral therapy for insomnia (CBT-I) and passive body heating (PBH) sessions using a sauna blanket over a 9-week treatment period to adults aged 18 years or older with insomnia disorder.

DETAILED DESCRIPTION:
Insomnia disorder is a common and consequential mental health problem, with prevalence estimates at approximately 10%. The American College of Physicians recommends cognitive behavioral therapy for insomnia (CBT-I), an efficacious "mind" (psychological and behavioral) treatment, as the first-line treatment for adults with insomnia. Yet, about half of individuals experience residual insomnia symptoms after CBT-I. Accordingly, researchers have sought to augment CBT-I, primarily with pharmacotherapy, but many people do not want to use pharmacologic agents due to concerns about side effects and dependence. Passive-body heating (PBH), a "body" treatment, involves heating the body via hot baths or showers, infrared sauna, or other heat sources. PBH has been found to reduce the time needed to fall asleep and to improve sleep quality. PBH may improve sleep by increasing skin temperature and decreasing core body temperature, a dynamic associated with sleep onset. CBT-I and PBH thus target distinct factors that may contribute to insomnia, and the investigators hypothesize that the combination of CBT-I and PBH holds promise as a multi-component treatment for insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Willing to use birth control if assigned female sex at birth
* Location to plug sauna blanket into regular wall outlet
* Ability to lie in sauna blanket for 15 minutes
* Ability to fit in the sauna blanket (no taller than 6' 3", no greater than 250 lbs)
* Daily access to the internet via computer, smartphone, or tablet
* Elevated insomnia symptoms as indexed by a score of 11 or greater on the Insomnia Severity Index (ISI)
* Insomnia disorder (characterized by difficulty initiating sleep) as indexed by a positive diagnosis on the Structured Clinical Interview for DSM-5 Sleep Disorders (SCISD)

Exclusion Criteria:

* Night shift worker
* Current or planned routine body heating practices (e.g., saunas, hot tubs)
* Pregnant or plans to become pregnant during the participation period
* Other diagnosed sleep disorders or suspected sleep disorders
* Medical conditions that might increase the risk of passive body heating using an infrared sauna blanket
* Mental health disorder that may better explain insomnia, require priority treatment, or be exacerbated by time in bed restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 9 weeks
  Proportion of eligible prospective participants who consent to complete at least 6 weeks of at least 3 PBH sessions per week over the 9-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final IPD dataset will include self-reported demographic data, other self-reported data (e.g., subjective sleep measures, mood symptoms), and wearable-derived sleep data (wearable-derived sleep data will be shared as nightly aggregates).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months after the publication of results and unending.
Access Criteria: Data will be accessible via the Vivli platform. To access IPD arising from this project, users must complete the Vivli data request form and sign the Vivli Data Use Agreement, which limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to reidentify research participants or engage in any unauthorized uses of the data. In order to get access to the data, the user must submit a valid scientific question, include a statistical analysis plan, and complete all required fields on the Vivli data request form. Vivli will review the data request for completeness. Anyone who has submitted an approved data request and signed a data use agreement on Vivli will be given access to the data. Vivli will then make the data available, without cost, to users for a set period of time. Vivli will maintain storage and access of the data for as long as it maintains scientific utility.
URL: https://vivli.org

REFERENCES:
- [Background] Lee S, Oh JW, Park KM, Lee S, Lee E. Digital cognitive behavioral therapy for insomnia on depression and anxiety: a systematic review and meta-analysis. NPJ Digit Med. 2023 Mar 25;6(1):52. doi: 10.1038/s41746-023-00800-3. PMID 36966184
- [Background] Haghayegh S, Khoshnevis S, Smolensky MH, Diller KR, Castriotta RJ. Before-bedtime passive body heating by warm shower or bath to improve sleep: A systematic review and meta-analysis. Sleep Med Rev. 2019 Aug;46:124-135. doi: 10.1016/j.smrv.2019.04.008. Epub 2019 Apr 19. PMID 31102877